CLINICAL TRIAL: NCT03112837
Title: Effect of Live Combined Bifidobacterium,Lactobacillus and Enterococcus Capsules on Oral Mucositis in Nasopharyngeal Carcinoma Patients Receiving Radiotherapy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Qiang Xu, head of Science and Euducation Division, Jiangxi Provincial Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: yjcl2017
Record Dates: First submitted 2017-03-31; First posted 2017-04-13 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Oral Mucositis; Quality of Life
MeSH Terms: conditions — Stomatitis | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- drug group (Experimental): live Lactobacillus, Bifidobacterium and Enterococcus ( two pills two times a day)with radiotherapy and Chemotherapy
  Interventions: Other: Lactobacillus, Bifidobacterium and Enterococcus
- non-drug group (No Intervention): only receiving radiotherapy and chemotherapy
- healthy control group (No Intervention)

INTERVENTIONS:
Other: Lactobacillus, Bifidobacterium and Enterococcus — 3 pills two times a day during the whole treatment
  Arms: drug group

SUMMARY:
Effect of Live Combined Bifidobacterium,Lactobacillus and Enterococcus Capsules on Oral Mucositis in Nasopharyngeal Carcinoma Patients Receiving Radiotherapy.

DETAILED DESCRIPTION:
Radiation-induced mucositis is an acute reaction of the mucosa of patients undergoing head and neck radiotherapy.It can lead to dose-limiting and debilitating side effect. There is no guideline on an acknowledged intervention that significantly reduces its severity. In the mucosa, the immune system's T cells and B cells have position-specific phenotypes and functions that are influenced by the microbiota. These cells play pivotal parts in the maintenance of immune homeostasis by suppressing responses to harmless antigens and by enforcing the integrity of the barrier functions of the gut mucosa.We designed a randomized trial of Live Combined Bifidobacterium,Lactobacillus and Enterococcus Capsules in patients with Nasopharyngeal Carcinoma. The aim of this study was to determine if regulating intestinal tract flora was effective in reducing the severity of radiation-induced mucositis in patients receiving radical dose radiotherapy. The effect of this intervention on a patient's general well-being was also investigated. The primary end-point of the study was the incidence of Radiation Therapy Oncology Group grade 3 mucositis.In 2017, 40 patients are estimated to be recruited into the study at Jiangxi Cancer Hospitals, China.20 patients were randomized to receive Live Combined Bifidobacterium,Lactobacillus and Enterococcus Capsules and 20 to receive a placebo.

ELIGIBILITY:
Inclusion Criteria:

Karnofsky score ≥80 newly diagnosed NPC without distant metastasis confirmed by pathology without any other malignant disease history no any other anti-cancer treatment for NPC previously received radiotherapy and chemotherapy at our Cancer Center

Exclusion Criteria:

any immune system disease under high risk to antimicrobial agents such as Diabetes,infection disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-01-05 (Estimated); Study Completion 2018-01-05 (Estimated)

PRIMARY OUTCOMES:
the incidence of Radiation Therapy Oncology Group grade 3 mucositis | one year
  confluent pseudomembranous mucosa

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, MD PHD, Principal Investigator — Jiangxi Provincial Cancer Hospital
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xia C, Jiang C, Li W, Wei J, Hong H, Li J, Feng L, Wei H, Xin H, Chen T. A Phase II Randomized Clinical Trial and Mechanistic Studies Using Improved Probiotics to Prevent Oral Mucositis Induced by Concurrent Radiotherapy and Chemotherapy in Nasopharyngeal Carcinoma. Front Immunol. 2021 Mar 24;12:618150. doi: 10.3389/fimmu.2021.618150. eCollection 2021. PMID 33841399